CLINICAL TRIAL: NCT00416234
Title: Laparoendoscopic Rendez Vous (Intraoperative ERCP) vs Two Stage Approach (Preoperative ERCP Followed by Laparoscopic Cholecystectomy) for the Management of Cholelithiasis/Choledocholithiasis
Brief Title: Laparoendoscopic Rendez Vous Versus Standard Two Stage Approach for the Management of Cholelithiasis/Choledocholithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Thessaly (Other)
Collaborators: Larissa University Hospital (Other)
Responsible Party: George Tzovaras, MD, University of Thessaly, School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Larissa CBD stones trial
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Last update posted 2010-01-14 (Estimated); Status verified 2008-06

CONDITIONS: Choledocholithiasis; Cholelithiasis
MeSH Terms: conditions — Choledocholithiasis; Cholelithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Laparoendoscopic Rendez vous (one stage management of cholelithiasis/choledocholithiasis)
  Interventions: Procedure: Laparoendoscopic Rendez vous
- 2 (Active Comparator): preoperative ERCP and CBD clearance followed by lap cholecystectomy (two stage management of cholelithiasis/choledocholithiasis)
  Interventions: Procedure: preoperative ERCP and CBD clearance

INTERVENTIONS:
Procedure: Laparoendoscopic Rendez vous — intraoperative ERCP for CBD clearance during laparoscopic cholecystectomy
  Arms: 1
Procedure: preoperative ERCP and CBD clearance — ERCP and CBD clearance followed by laparoscopic cholecystectomy
  Arms: 2

SUMMARY:
The purpose of the study is to assess whether combined intraoperative ERCP and CBD clearance with laparo-endoscopic rendez-vous during laparoscopic cholecystectomy (one stage approach) is or not superior to the standard practice of preoperative ERCP, sphincterotomy and CBD clearance followed by laparoscopic cholecystectomy (two stage approach) in patients with combined cholelithiasis and choledocholithiasis.

DETAILED DESCRIPTION:
The ideal management of concomitant cholelithiasis and choledocholithiasis is not known yet. There are several options, including one-stage or two-stage approaches. The most commonly used practice is the two-stage management which consists of preoperative ERCP, sphincterotomy and CBD clearance followed by laparoscopic cholecystectomy. However, with this approach, a number of patients will be submitted to an unnecessary ERCP while some others will develop complications, mainly pancreatitis due to inadvertent pancreatic duct cannulation. Laparo-endoscopic rendez-vous methods have been described in order to obtain selective CBD cannulation and omit the risk of post-ERCP pancreatitis. In this procedure, during laparoscopic cholecystectomy, a wire is inserted through the cystic duct into the common bile duct, advanced into the duodenum where is found endoscopically, gripped with a snare and retrieved through the mouth. The a sphincterotome is inserted over the wire and elective CBD cannulation is obtained to be followed by sphincterotomy and CBD clearance intraoperatively. The method has been described by several authors in small to moderate case series, its safety has been proven and it appears that reduces both the length of hospital stay and the incidence of post-ERCP pancreatitis.However, it has not been popularized and has never been tested over the standard two-stage management. In our hospital, the standard approach for cholelithiasis and choledocholithiasis has been, as well, the two-stage (preop ERCP and sphincterotomy followed by laparoscopic cholecystectomy)approach. We initially assessed the feasibility and safety of the laparo-endoscopic rendez vous with a pilot study and now we intend to compare the two methods in a prospective randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* patients must be able to give informed consent preoperatively
* ASA I-III
* patients at high risk to have CBD stones (jaundice, cholangitis, grossly deranged LFTs, CBD stones found on US or MRCP)

Exclusion Criteria:

* patients not fit for surgery (ASA IV)
* previous ERCP and sphincterotomy
* previous upper abdominal surgery
* pregnancy at time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-09; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
postoperative hospital stay | from onset of intervention to discharge

SECONDARY OUTCOMES:
success rate of CBD clearance | during ERCP
failure rate of selective CBD cannulation | during ERCP
incidence of multiple endoscopic procedures | within 30 days
incidence of hyperamylasemia | within 48 hours post-ERCP
incidence of severe pancreatitis (APACHE II score >6) | within 48 hours post-ERCP
total hospital stay | from admission to discharge
complications other but pancreatitis | within 30 days
death | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Hatzitheofilou, MD, Study Chair — University of Thessaly, School of Medicine; George Tzovaras, MD, Study Director — University of Thessaly, School of Medicine; Ioannis Baloyiannis, MD, Principal Investigator — University Hospital of Larissa
Locations (1):
- University Hospital of Larissa, Larissa, Thessaly, Greece

REFERENCES:
- [Derived] Tzovaras G, Baloyiannis I, Zachari E, Symeonidis D, Zacharoulis D, Kapsoritakis A, Paroutoglou G, Potamianos S. Laparoendoscopic rendezvous versus preoperative ERCP and laparoscopic cholecystectomy for the management of cholecysto-choledocholithiasis: interim analysis of a controlled randomized trial. Ann Surg. 2012 Mar;255(3):435-9. doi: 10.1097/SLA.0b013e3182456ec0. PMID 22261836